CLINICAL TRIAL: NCT06776302
Title: Assessment of Brain Damage Using Monitoring of Cerebral Oximetry Dynamics in Patients After Cardiac Arrest
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Maribor (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UKC Maribor OIIM/UC/KN
Record Dates: First submitted 2025-01-09; First posted 2025-01-15 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Cardiac Arrest (CA)
Keywords: cardiac arrest, near infrared spectroscopy
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients after cardiac arrest (Experimental): Patients after cardiac arrest, admited to department of Intensive internal medicine.
  Interventions: Diagnostic Test: Raise of blood flow through the brain

INTERVENTIONS:
Diagnostic Test: Raise of blood flow through the brain — At each patient two test are preformed. The first test is based on increasing blood flow through the brain through a controlled gradual infusion of norepinephrine (noradrenalin). The patient will receive such an infusion immediately upon admission and stabilization in the Department of Intensive Internal Medicine and then in the period of 6, 12, 24, 48 and 72 hours after admission. The second test is based on passive elevation of the lower extremities. The second test will also be performed on the patient immediately upon admission and stabilization in the Department of Intensive Internal Medicine and then in the period of 6, 12, 24, 48 and 72 hours after admission.

SUMMARY:
Sudden cardiac arrest is one of the leading causes of death in Europe. The recommended treatment for cardiac arrest is cardiopulmonary resuscitation (CPR) and electrical defibrillation with an automated external defibrillator (AED).

The chain of survival, which connects all links of basic and additional resuscitation procedures and post-resuscitation care, is important for successful survival.

Most patients after out-of-hospital cardiac arrest die in intensive care units due to the withdrawal of active treatment, based on the prediction of a poor neurological outcome. Prognostic indicators are influenced by many factors, including the patient's neurological condition. This should be taken into account when predicting outcome and a multimodal approach based on clinical examination, electrophysiological examinations, imaging studies and biological markers should be used.

Based on the professional literature, we asked ourselves the research question of whether it is possible to achieve changes in cerebral oxygen saturation values using simple tests and whether such changes in cerebral oxygen saturation coincide with other methods used to assess neurological outcome and brain damage in patients after primary out-of-hospital cardiac arrest. The patient will have a device installed to detect cerebral oxygen saturation (NIRS) throughout the entire hospitalization period. The level of oxygen in the brain is influenced by various factors: mean arterial pressure, cardiac index, carbon dioxide level in the blood, hemoglobin level in the blood, depth of sedation, body temperature. We will attempt to achieve changes in cerebral oxygen saturation with two simple tests. The first test is based on increasing blood flow through the brain through a controlled gradual infusion of a drug that raises blood pressure. The patient will receive such an infusion immediately upon admission and stabilization in the Department of Intensive Internal Medicine and then in the period of 6, 12, 24, 48 and 72 hours after admission.

The second test is based on passive elevation of the lower extremities, which results in a transient increased cardiac index produced by the heart and a consequent increase in blood flow through the brain. The second test will also be performed on the patient immediately upon admission and stabilization in the Department of Intensive Internal Medicine and then in the period of 6, 12, 24, 48 and 72 hours after admission.

Based on the data obtained with the help of the aforementioned tests, we will not decide on the prognosis of the patient's neurological outcome or change or adjust the therapy in any way based on the data obtained.

The aim of the study is to demonstrate that changes in cerebral oxygen saturation values in patients after primary out-of-hospital cardiac arrest, obtained with simple tests, coincide with other methods used to assess neurological outcome and brain damage.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Primary out-of-hospital cardiac arrest
* Unconsciousness after return of spontaneous circulation (8 points or less on the Glasgow Coma Scale)

Exclusion Criteria:

* Intracranial hemorrhage (clinically suspected or proven by CT scan)
* Hypothermia (body temperature less than 32 degrees Celsius)
* Pregnancy
* Uncontrollable bleeding
* Uncontrollable blood pressure fluctuations
* Patient defined as palliative or terminal
* Cardiac arrest secondary to drowning, hypothermia, or trauma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Changes in cerebral oximetry values in patients after primary out-of-hospital cardiac arrest, obtained with described tests | From enrollment to the 2 days after admission

CONTACTS AND LOCATIONS:
Locations (1):
- University clinical center Maribor, Maribor, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided